CLINICAL TRIAL: NCT04299230
Title: Continous Monitoring of Vital Signs on Hospitalized Cancer Patients.
Acronym: InnoCan WP4
Status: Completed | Type: Observational
Sponsor: Naestved Hospital (Other)
Responsible Party: Principal Investigator, Niels Henrik Holländer, Head of Department, MD, Naestved Hospital
Other Study IDs: COR 20151
Record Dates: First submitted 2016-02-16; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Cancer; Fever
Keywords: Febrile hospitalized cancer patients
MeSH Terms: conditions — Neoplasms; Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cortium C3

SUMMARY:
Clinical Data Validation of a Novel Continuous Vital Sign Monitoring System in Cancer Patients Background The Cortrium C3 device is a novel, inexpensive, chest-worn unit designed for measuring vital sign parameters. The unit is capable of logging and wireless transmitting data describing pulse, respiratory rate, body surface temperature, ambient temperature and accelerometer data (1,2). The C3 device is developed as a diagnostic tool in the medical practice to meet the demand for a modern reliable and open medical grad vital sign monitoring system. The device is based on state-of-the-art technologies and is produced using high quality off-the-shelf components. Although, new technologies may be of high value to the health care system, studies show that the quality of technologies vary and more empiric data is needed to either support or reject the advantages of using intelligent health technologies at home (3-5). Besides measuring the actual quality of C3, it is therefore also important to evaluate how patients experience quality in relation to C3 in addition to an evaluation of perspectives from the health professionals.

Objective The objective of the study is to validate measurements of pulse, frequency of respiration, and temperature obtained with the C3 device by comparison with routinely used hospital equipment. Further, the objective is to gain knowledge about how patients experience to be monitored with C3 and how hospital staff experience working with C3.

Design and participants The study is carried out on cancer patients at the Department of Oncology, Naestved Hospital, Region Zealand, Denmark (DONZ). Collaborating partners are Cortrium, University College Zealand and Sundhedsinnovation Zealand.

The study consists of a quantitative and a qualitative part. The quantitative study is a cross-sectional study of paired measures of vital sign parameters (pulse, respiratory rate and temperature) measured by the C3 device and standard hospital equipment used at DONZ. The qualitative study is planned as observational studies and semi-structured interviews with patients, who have been monitored with C3 and health professionals who have been involved in treatment or care of monitored patients. Recruitment of participants will take place amongst newly hospitalized patients at DONZ. It is planned to include approximately 40 patients in February and March 2016.

Side effects, risks and inconveniences No major side effects are related to wearing and being monitored by the C3 device. The device has been tested on healthy volunteers and reports of inconveniences are mostly related to the adhesive ECG-electrodes that can irritate the skin. However, a wide array of electrodes are commercially available to fit the individual needs. Some might find wearing the device stigmatizing and/or inconvenient.

In addition, the C3 device is marked CE class I. Hence, requirements for prevention of adverse effects are met. As an example, this includes two fuses between the battery and the electrodes, minimizing the risk of current for the battery entering the body even in the event of device failure. The device has not yet been approved for commercialization.

Ethics and anonymization All data collected in the study is done according to the guidelines of Good Clinical Practice (GCP) for medical device studies (6). All data is anonymized, and is protected according to national law: "Lov om behandling af personoplysninger". The project has been reported to "Datatilsynet" [the Data Protection Agency].

Test subjects are secured access to further information about the study through their assigned nurse or email and telephone.

Approvals The study has been approved by the Danish Ethical Comity: SJ-460, and The Danish Medicines Agency: journal number 2015120113.

DETAILED DESCRIPTION:
Clinical Data Validation of a Novel Continuous Vital Sign Monitoring System in Cancer Patients

Background The Cortrium C3 device is a novel, inexpensive, chest-worn unit designed for measuring vital sign parameters. The unit is capable of logging and wireless transmitting data describing pulse (electrocardiogram), respiratory rate, body surface temperature, ambient temperature and accelerometer data. The C3 device is developed as a diagnostic tool in the medical practice to meet the demand for a modern reliable, and open medical grad vital sign monitoring system. The device is based on state-of-the-art technologies and is produced using high quality off-the-shelf components.

In Denmark, 80 % of the total health finances are used to treat and care for persons with chronical diseases. The number of chronically ill citizen is increasing, and at the same time the demographic development implies an increasingly older population (1). New health technologies are seen as one of the future solutions of economic and demographic challenges of the healthcare system. In addition, continuously wireless monitoring of ill patients at home or in a clinical setting may facilitate early detection of critical development of vital signs in patients. Thus, it is believed that introduction of new smart and wireless technologies will affect and alter todays manually performed gold standard methods of measuring vital sign parameters. The C3 device is such a technology.

The patients participating in the project are cancer patients in the Department of Oncology, Naestved Hospital, Region Zealand, Denmark. The cancer patients affiliated to the Department are monitoring body temperature at home, and it is often fever (> 38,5 ° C) that is the cause of hospitalization. Thus, continuously measurement of the temperature at home by the C3 device could be helpful in detection of temperature rise. However, in the literature surface temperature above sternum has not been correlated to core temperature. In fact, no direct association between surface temperature and body temperature has been described in the literature. However, a review from 2014 addresses a number of considerations about the relation between surface temperature and body temperature (2). Thus, the evaluation of surface and ambient temperature measured by C3 in comparison with clinically measure temperature in the present study will be of explorative nature.

Although, new technologies may be of high value to the health care system, studies show that the quality of technologies vary and more empiric data is needed to either support or reject the advantages of using intelligent health technologies in the home (3-5). Besides measuring the actual quality of C3, it is therefore also important to evaluate how patients experience quality in relation to C3 in addition to an evaluation of perspectives from the health professionals.

Brief overview of technical specifications of C3 Table 1 display an overview of the vital parameters measured by the C3 device in the present study. Further, an accelerometer is embedded enabling various medically relevant derived measures, which will not be evaluated in the present study. The C3 device is attached directly above the sternum using standard electrodes

Pulse / heart rate C3 heart rate measurement is derived from QRS-complex detection in the ECG signal using an existing open source algorithm (6). Under normal cardiovascular circumstances the peripheral pulse and ECG-derived heart rate is assumed to be identical.

Respiratory rate Respiratory rate measured by the C3 device is impedance-based. This implies that the signal changes are based on changes in the electrical resistance of the alternating current circuitry. Impedance is increased due to the following two effects: 1) During inspiration there is an increase of the gas volume of the chest in relation to the fluid volume. This increase causes conductivity to decrease. 2) During inspiration, the length of the conductance paths increases because of expansion.

There is a good correlation between this impedance change and the volume of inhaled. This relationship is linear (7).

Temperature C3 measures body surface on the torso directly above the sternum. The sensor is an infrared optical thermometer with a specified accuracy of ± 0.2 ℃. Further, the C3 device measures ambient temperature with a thermometer embedded into the printed circuit board. There is no evidence found in the literature about a correlation between body surface temperature and body core temperature.

Objective The objective of the study is to validate measurements of pulse, frequency of respiration, and temperature obtained with the C3 device by comparison with routinely used hospital equipment. Further, the objective is to gain knowledge about how patients experience to be monitored with C3 and how hospital staff (primarily nurses) experience working with C3.

Participants and design The study consists of a quantitative and a qualitative part. The quantitative study is a cross-sectional study of paired measures of vital sign parameters (pulse, respiratory rate and temperature) measured by C3 and standard hospital equipment used at the Department of Oncology, Naestved Hospital. The qualitative study is planned as observational studies and semi-structured interviews with patients, who have been monitored with C3 and health professionals who have been involved in treatment or care of monitored patients. Recruitment of participants will take place amongst newly hospitalized patients at the Department of Oncology, Naestved Hospital. It is planned to include approximately 40 patients in February and March 2016. A total of ten C3 devices and their corresponding tablets will be included in the study.

Inclusions criteria Legally competent persons age 18 or older with a cancer diagnosis, who are enrolled at the Department of Oncology, Naestved Hospital and who are febrile (> 38,5 °C). Exclusion criteria Pregnant and fertile women, who does not use contraceptives. Patients with known heart disease.

Informed consent Patients will upon hospitalization receive verbal and written information about the study. Patient who agree to participate sign a declaration of informed consent. Since the aim of the study is to evaluate vital parameters in the acute face, patients are asked to give informed consent during the first 24 hrs. If patients are hospitalized during the night shift information about the study will be given in the first day shift after hospitalization.

Method The study initiates when the patient has given informed consent, after which the C3 device is placed on the patient. Following this the patients will be monitored according to the current clinical guidelines at Department of Oncology, Naestved Hospital. When clinical assessment of vital parameters is terminated, the C3 device is removed. This will most often be at the end of hospitalization.

Quantitative design Paired measures of vital parameters measured by C3 and by hospital equipment currently used at Department of Oncology, Naestved Hospital will be compared.

All patients at Department of Oncology, Naestved Hospital are risk assessed upon hospital admission. Patients are scored from 0-3 points in each parameter (higher is worse). Future and/or acute action is based on changes in individual parameters or accumulated score. Measurements are done by nurses and either measured using medical equipment or assessed manually. Values are handwritten on a risk-assessment-sheet before being entered into the local electronic patient care system (Opus). Time of registration and room temperature will additionally be registered.

Inpatients are risk-assessed at least three times during the first 24 hours of their hospital stay. Subsequent risk-assessment interval is based on risk-score, and will take place at least once every 24 hours until hospital discharge.

A research nurse will several times a week transfer the manually registered data and time-identical data from the C3 device into an anonymized data sheet. Additionally, information about gender, age, weight, height and diagnoses will be withdrawn from the patient journals and registered in the anonymized data sheet. Registrations will continue during the entire hospital admission.

The staff of the department will continue their daily routines, and will only be involved in recruitment of possible participants and the placement/removal and daily recharging of the C3 device.

Upon removal, the C3 device will be cleaned and disinfected according to the hygiene regulations of the department.

No biological material is sampled from patients and no biobank is created.

Statistical considerations Statistical analysis of measurements for data validation is done using Bland-Altman plots (difference plots) which allows for investigation of the existence of any systematic difference between the measurements and to identify possible outliers. The recommended 95% limits of agreement (mean difference plus or minus 1.96 standard deviations) will be used, which would give information about how far apart measurements by the two methods are likely to be for most individuals. If the differences within mean ± 1.96 SD are not clinically important, the two methods may be used interchangeably (8-10). Accordingly, estimates (confidence intervals) for "limits of agreement" will be calculated.

In method-comparison studies, increasing the number of paired measurements is pivotal. This number will determine the limits of agreement (confidence interval). A sample of 200 paired measurements (n=200) yields a 95% CI about +/- 0.24s. Hence this is the target number of measurements to reach.

Number of patients: The aim is to carry out 200 paired measurements. Since the study includes ten C3 devices it is calculated, that on average each device shall provide twenty registrations. Since vital parameters will be registered at least once a day in patients hospitalized in Department of Oncology, Naestved Hospital it will take a total of at least twenty days to obtain the required number of measurements. The project period is planned to be seven weeks. The Department have approximately 22-28 new admissions per week with an approximate admission time of 5,4 days. This means that in 49 days (seven weeks) a total of approximately 90 patients (49 days/5,4 days * 10 C3 devices) will be available for the recruitment procedure. In this population it is expected that 60 % is hospitalized with a temperature above 38,5 °C and therefore meet the inclusion criteria. Dropout is estimated to 25 %, which results in an estimated total population of approximately 40 patients. However, the demand of 200 paired measurements will be determining the final number of patients included in the study.

Qualitative design Interviews: The purpose of the qualitative part of the study is to investigate 1) how patients experience to wear an being continuously monitored with the C3 device, and 2) what challenges health professionals experience in their work, when patients are wearing the C3 device.

The qualitative part of the study is based on semi-structured interviews with twelve participating patients during their hospital admission. In addition, ten health professionals who have been involved in treatment and care of patients wearing the C3 device will be interviewed.

Observation: Observational studies are carried out to elucidate possible challenges related to treat and care patients that are wearing the C3 device. The observational studies will be are carried out before making the semi-structured interviews, so observations can qualify the questions asked in the interviews.

Side effects, risks and inconveniences No major side effects are related to wearing and being monitored by the C3 device. The device has been tested on healthy volunteers and reports of inconveniences are mostly related to the adhesive ECG-electrodes that can be painful to remove and/or irritate the skin. However, a wide array of electrodes are commercially available to fit the individual needs (e.g., sensitive skin or allergy). Some might find wearing the device stigmatizing and/or inconvenient.

In addition, the C3 device is marked CE class I. Hence, requirements for prevention of adverse effects are met. As an example, this includes two fuses between the battery and the electrodes, minimizing the risk of current for the battery entering the body even in the event of device failure. The device has not yet been approved for commercialization.

Ethics and anonymization All data collected in the study is done according to the guidelines of Good Clinical Practice (GCP) for medical device studies (11). All data is anonymized, and all data is protected according to national law: "Lov om behandling af personoplysninger". The project has been reported to "Datatilsynet" [the Data Protection Agency].

Test subjects are secured access to further information about the study through their assigned nurse or email and telephone (contact information is in the information material).

Economics The responsible researchers are not economically compensated for the work in this study. Participating patients do not receive compensation for their participation.

Publications At least one scientific paper will be published upon completion of the study.

Approvals The study has been approved by the Danish Ethical Comity (Region Zealand): SJ-460, and The Danish Medicines Agency: journal number 2015120113.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized febrile cancer patient. Temperatur above 38,5 C -
* 18 years old or more

Exclusion Criteria:

* Fertile women, not using birth control
* Pregnant women
* Inhabile patient, not able to understand information -
* Known heaert disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized febrile cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Comparing vital sign parameters of temperature, pulse and respiratory rate from C3 device with manual nurse registration | 24 months
  Comparing data fra C3 device with the data collected by standard hospital equipment used at the Department of Oncology

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Naestved Hospital, Næstved
  - Næstved